CLINICAL TRIAL: NCT04426656
Title: IGHID 12001 - The Development of a Mobile-based App to Increase Uptake of Pre-Exposure Prophylaxis (PrEP) by Men Who Have Sex With Men in China
Brief Title: The Development of a Mobile-based App to Increase Uptake of Pre-Exposure Prophylaxis (PrEP) by Men Who Have Sex With Men in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-3481; R01AI114310 (NIH)
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-01

CONDITIONS: HIV; Pre-exposure Prophylaxis
Keywords: HIV; PrEP

STUDY DESIGN:
Intervention Model Description: Mixed methods study, including a 2-arm randomized controlled trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 2 Standard of Care (No Intervention): Participants will receive written HIV prevention materials including basic facts of PrEP, recommendations for HIV/STI(sexually transmitted infections) testing and referrals to local HIV/STI testing sites and prevention services.
- Part 2 mini-app (Experimental): In addition to the standard of care, participants in the mini-app arm will have access to the mini-app (i.e. the intervention) during the whole study period.
  Interventions: Behavioral: Phone application

INTERVENTIONS:
Behavioral: Phone application — The mini-app (used in Part 2) has four main functions:
  1. a knowledge center that contains a series of HIV-, sexual health-, and PrEP-related educational articles in Chinese;
  2. an HIV self-test toolkit ordering system that allows users to order a finger-prick HIV rapid test toolkit and shipped to home for free (one piece at a time);
  3. an asynchronous message function that allows users to chat with a study staff (C.Li); and
  4. a user profile page where users can manage all HIV test orders.
  Other Names: mini-app
  Arms: Part 2 mini-app

SUMMARY:
This study aims to use a mini-application on the popular Chinese social media mobile platform, WeChat, to improve HIV pre-exposure prophylaxis (PrEP) uptake among at-risk men who have sex with men (MSM). UNC investigators will work in close partnership with a well-established HIV special hospital and the local MSM community to understand key barriers to PrEP use, and develop a mobile-based intervention to increase PrEP uptake among young MSM in Guangzhou, China.

DETAILED DESCRIPTION:
This study includes two parts. Before the start of Part 1, a mini-app prototype for promoting HIV pre-exposure prophylaxis (PrEP) uptake will have been developed from a prior MSM community-driven hackathon contest. PrEP is an antiretroviral medicines-based prevention strategy against HIV infection, which has been proved save and effective.

Part 1 includes in-depth interviews with 40 HIV-negative young MSM (18 and above) with a brief survey to collect demographic data. The interview topics include PrEP-related perceptions and feedback on the design of a mini-app prototype. Findings from Part 1 will inform refining the mini-app before the start of Part 2.

In Part 2, a small two-arm randomized control trial with 70 young MSM (18 and above) will be conducted to evaluate the preliminary efficacy of the mini-app in improving PrEP-related perceptions and actual PrEP uptake, compared to a control group of standard of care.

Participants in Part 2 will be followed up for 12 weeks (8 week intervention and after-intervention follow-up at 12th week). A subgroup of participants (n=15) from both the intervention arm and the control arm will receive two rounds of in-depth interviews, separately at the 4th and 8th week, to share their experience of using the app and changed perceptions and/or behaviors related to PrEP.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: HIV-negative men who have sex with men (MSM): must self-report: being assigned male sex at birth, HIV-negative, age 18 and above, ever having had anal sex with another man, identify as a Chinese citizen, own a smartphone, able to being willing to sign written informed consent and participate in the study as procedures required.

Part 2: HIV-negative men who have sex with men (MSM): same characteristics as in Part 1.

AND, they must report :

* Having a smartphone with WeChat installed.
* Being assigned male sex at birth, HIV-negative, age 18 and above, ever having had anal sex with another man, currently reside in Guangzhou, China, identifying as a Chinese citizen, able to sign written informed consent and participate in the study as procedures require. AND
* At least one criterion associated with high risk of HIV infection in the past 6 months prior to enrollment as follows:

  * Unprotected (condomless) anal intercourse with male partner(s)
  * More than two male partners (regardless of condom use and HIV serostatus)
  * Reported STI, such as syphilis, Herpes Simplex Virus-2 (HSV-2), gonorrhea, chlamydia, chancroid, or lymphogranuloma venereum.
  * Reported use of post-exposure prophylaxis (PEP)
  * Have a sexual partner living with HIV

Exclusion Criteria:

* Part 1: Individuals who report any following status will be excluded from participating Part 1:

  * HIV-positive
  * Mental health issues which may compromise participant adherence or safety, including memory loss, cognitive impairment, intellectual disability, or communication disorders.
* Part 2:

  * HIV-positive (self-report or lab-confirmed)
  * Currently taking oral PrEP based on self-report
  * Symptoms of acute HIV infection within the prior 30 days
  * Contradictions to taking oral PrEP
  * Personal diagnosis or family history of hemophilia
  * Chronic Hepatitis B (self-report)
  * Participating in another research study related to HIV and antiretroviral therapy or other intervention study
  * Having serious chronic disease, including metabolic diseases (such as diabetes), neurological, and psychiatric disorders
  * Mental health issues which may compromise participant adherence or safety, including memory loss, cognitive impairment, intellectual disability, or communication disorders

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This is a tailored intervention pilot study for MSM in China
Enrollment: 70 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chunyan Li, MS, Principal Investigator — University of North Carolina; Joseph D Tucker, MD, Study Director — University of North Carolina
Locations (1):
- Guangzhou No. 8 People's Hospital, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: Beginning 9 and ending 36 months following article publication.
Access Criteria: Investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Li C, Xiong Y, Maman S, Matthews DD, Fisher EB, Tang W, Huang H, Mu T, Tong X, Yu J, Yang Z, Sherer R, Hazra A, Lio J, Li L, Tucker JD, Muessig KE. An instant messaging mobile phone application for promoting HIV pre-exposure prophylaxis uptake among Chinese gay, bisexual and other men who have sex with men: A mixed methods feasibility and piloting randomized controlled trial study. PLoS One. 2023 Nov 13;18(11):e0285036. doi: 10.1371/journal.pone.0285036. eCollection 2023. PMID 37956177
- [Derived] Li C, Xiong Y, Muessig KE, Tang W, Huang H, Mu T, Tong X, Yu J, Yang Z, Sherer R, Hazra A, Lio J, Matthews DD, Fisher EB, Li L, Tucker JD. Community-engaged mHealth intervention to increase uptake of HIV pre-exposure prophylaxis (PrEP) among gay, bisexual and other men who have sex with men in China: study protocol for a pilot randomised controlled trial. BMJ Open. 2022 May 10;12(5):e055899. doi: 10.1136/bmjopen-2021-055899. PMID 35537794

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 2 Standard of Care: Participants will receive written HIV prevention materials including basic facts of PrEP, recommendations for HIV/STIs testing and referrals to local HIV/STIs testing sites and prevention services.
- Part 2 Mini-app: In addition to the standard of care, participants in the mini-app arm will have access to the mini-app (i.e. the intervention) during the whole study period.
  Phone application: The mini-app (used in Part 2) has four main functions:
  1. a knowledge center that contains a series of HIV-, sexual health-, and PrEP-related educational articles in Chinese;
  2. an HIV self-test toolkit ordering system that allows users to order a finger-prick HIV rapid test toolkit and shipped to home for free (one piece at a time);
  3. an asynchronous message function that allows users to chat with a study staff (C.Li); and
  4. a user profile page where users can manage all HIV test orders.
Period: Overall Study
Arm/Group | Part 2 Standard of Care | Part 2 Mini-app
Started | 24 | 46
Completed | 21 | 43
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 2 Standard of Care | Part 2 Mini-app | Total
Number analyzed (Participants) | 24 | 46 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (4.6) | 28.2 (6.8) | 28.0 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 24 | 46 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 46 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 24 | 46 | 70
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 24 | 46 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change in Intention to Use PrEP Score
Description: Individual perceived likelihood to start using PrEP, measured by a one-item question with a bipolar response scale (-3 to 3). Higher score indicates higher intention to use.
Time Frame: Baseline and up to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 2 Standard of Care | Part 2 Mini-app
Number analyzed (Participants) | 21 | 43
score on a scale
  Baseline to Week 4 | 0.19 (1.72) | 0.00 (2.32)
  Baseline to Week 8 | 0.57 (2.62) | -0.09 (2.29)
  Baseline to Week 12 | 1.00 (2.59) | -0.40 (2.59)
Statistical Analysis 1: Comparison: Part 2 Standard of Care vs Part 2 Mini-app; The comparison was made using the outcome variable measured at Week 12; Test type: Superiority; p = 0.85, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Number of Participants Who Initiate PrEP by Week 8
Description: Individual's self-reported whether starting use of PrEP medication (binary: Yes/No)
Time Frame: Up to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Standard of Care | Part 2 Mini-app
Number analyzed (Participants) | 24 | 46
Participants | 5 | 8
Statistical Analysis 1: Comparison: Part 2 Standard of Care vs Part 2 Mini-app; Test type: Superiority; p = 0.72, Chi-squared

3. Primary Outcome: Number of Participants at Different Change Stages to PrEP Initiation at Baseline
Description: Individual's stages in the changing process towards starting using PrEP, which includes pre-contemplation (no interest in using PrEP), contemplation (interested in using PrEP but no action taken), preparation (plan to start PrEP and have taken initial actions), action (have started using PrEP), and maintenance (stay adherent to PrEP regimen). Each stage will be assessed by 1 or 2 questions (Yes/No) to determine which stage the individual is currently at.
Time Frame: Baseline
Population: Only participants with no missing data were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Standard of Care | Part 2 Mini-app
Number analyzed (Participants) | 21 | 43
Participants
  Pre-contemplation | 9 | 15
  Contemplation | 8 | 24
  Preparation | 4 | 4
  Action | 0 | 0
Statistical Analysis 1: Comparison: Part 2 Standard of Care vs Part 2 Mini-app; Test type: Superiority; p = 0.318, Fisher Exact

4. Primary Outcome: Number of Participants at Different Change Stages to PrEP Initiation at Week 4
Description: as for outcome 3
Time Frame: Week 4
Population: Only participants with no missing data were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Standard of Care | Part 2 Mini-app
Number analyzed (Participants) | 21 | 43
Participants
  Pre-contemplation | 10 | 15
  Contemplation | 5 | 12
  Preparation | 6 | 12
  Action | 0 | 4
Statistical Analysis 1: Comparison: Part 2 Standard of Care vs Part 2 Mini-app; Test type: Superiority; p = 0.527, Fisher Exact

5. Primary Outcome: Number of Participants at Different Change Stages to PrEP Initiation at Week 8
Description: as for outcome 3
Time Frame: Week 8
Population: Only participants with no missing data were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Standard of Care | Part 2 Mini-app
Number analyzed (Participants) | 21 | 43
Participants
  Pre-contemplation | 8 | 20
  Contemplation | 4 | 7
  Preparation | 4 | 8
  Action | 5 | 8
Statistical Analysis 1: Comparison: Part 2 Standard of Care vs Part 2 Mini-app; Test type: Superiority; p = 0.928, Fisher Exact

6. Primary Outcome: Number of Participants at Different Change Stages to PrEP Initiation at Week 12
Description: as for outcome 3
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Standard of Care | Part 2 Mini-app
Number analyzed (Participants) | 21 | 43
Participants
  Pre-contemplation | 8 | 17
  Contemplation | 3 | 11
  Preparation | 5 | 7
  Action | 5 | 8
Statistical Analysis 1: Comparison: Part 2 Standard of Care vs Part 2 Mini-app; Test type: Superiority; p = 0.678, Fisher Exact

7. Secondary Outcome: Change in PrEP Knowledge Score at Week 4, 8 and 12
Description: Individual's understanding of PrEP, measured by a 5-item True/False quiz. Values range from 0-5. Higher score indicates better PrEP knowledge.
Time Frame: Baseline and up to 12 weeks
Population: Participants analyzed here only include those with complete data at a certain follow-up week.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 2 Standard of Care | Part 2 Mini-app
Number analyzed (Participants) | 21 | 43
score on a scale
  Baseline to Week 4 | 0.33 (0.72) | 0.13 (0.79)
  Baseline to Week 8 | 0.33 (0.66) | 0.16 (0.78)
  Baseline to Week 12 | 0.38 (0.50) | 0.19 (0.82)
Statistical Analysis 1: Comparison: Part 2 Standard of Care vs Part 2 Mini-app; The comparison test was made using the outcome variable measured at Week 12; Test type: Superiority; p = 0.26, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Number of Participants Who Are Willing to Pay a Specified Percentage of Monthly Income for PrEP
Description: Willingness to pay for PrEP ranging from 0-100% of monthly income. Amount spent will be assessed at Baseline, Weeks 4, 8, and 12.
Time Frame: Up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Standard of Care | Part 2 Mini-app
Number analyzed (Participants) | 21 | 43
Participants
  Baseline: Any amount | 0 | 6
  Baseline: 30-50% | 0 | 0
  Baseline: 15-25% | 0 | 4
  Baseline: 10-15% | 1 | 6
  Baseline: < 10% | 4 | 14
  Baseline: Not any | 9 | 5
  Baseline: Not sure | 3 | 4
  Baseline: Other | 4 | 4
  Week 4: Any amount | 0 | 4
  Week 4: 30-50% | 0 | 0
  Week 4: 15-25% | 0 | 7
  Week 4: 10-15% | 5 | 5
  Week 4: < 10% | 11 | 14
  Week 4: Not any | 1 | 7
  Week 4: Not sure | 1 | 3
  Week 4: Other | 3 | 3
  Week 8: Any amount | 0 | 5
  Week 8: 30-50% | 0 | 1
  Week 8: 15-25% | 1 | 4
  Week 8: 10-15% | 4 | 5
  Week 8: < 10% | 9 | 17
  Week 8: Not any | 2 | 6
  Week 8: Not sure | 3 | 3
  Week 8: Other | 2 | 2
  Week 12: Any amount | 0 | 3
  Week 12: 30-50% | 0 | 1
  Week 12: 15-25% | 2 | 5
  Week 12: 10-15% | 8 | 8
  Week 12: < 10% | 5 | 20
  Week 12: Not any | 2 | 4
  Week 12: Not sure | 1 | 2
  Week 12: Other | 3 | 0
Statistical Analysis 1: Comparison: Part 2 Standard of Care vs Part 2 Mini-app; The comparison was made using data measured at Week 12; Test type: Superiority; p = 0.08, Fisher Exact

9. Secondary Outcome: Change in PrEP Self-Efficacy Score
Description: Self-Efficacy will be assessed at Baseline, Weeks 4, 8, and 12 using an 8-item PrEP self-efficacy scale. Values range from 0-5. Higher scores indicate higher self-efficacy to use PrEP.
Time Frame: Baseline and up to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 2 Standard of Care | Part 2 Mini-app
Number analyzed (Participants) | 21 | 43
score on a scale
  Baseline to Week 4 | 0.05 (0.40) | 0.07 (0.39)
  Baseline to Week 8 | 0.08 (0.50) | 0.03 (0.41)
  Baseline to Week 12 | 0.10 (0.47) | 0.13 (0.44)
Statistical Analysis 1: Comparison: Part 2 Standard of Care vs Part 2 Mini-app; The comparison was made using data measured at Week 12; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Change in PrEP Attitude Score
Description: Individual's attitude towards PrEP, measured by a 5-item scale. Values range from 0-5. Higher scores indicate more positive attitude toward PrEP. The PrEP Attitude will be assessed at Baseline, Weeks 4, 8, and 12.
Time Frame: Baseline and up to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 2 Standard of Care | Part 2 Mini-app
Number analyzed (Participants) | 21 | 43
score on a scale
  Baseline to Week 4 | 0.06 (0.32) | 0.07 (0.66)
  Baseline to Week 8 | 0.23 (0.79) | 0.01 (0.72)
  Baseline to Week 12 | 0.02 (0.44) | 0.02 (0.72)
Statistical Analysis 1: Comparison: Part 2 Standard of Care vs Part 2 Mini-app; This comparison was made using data at Week 12; Test type: Superiority; p = 0.58, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Change in PrEP Stigma Score
Description: Individual's perceived stigma related to PrEP, measured by 5-item PrEP stigma scale. Values range from 0-5. Higher score indicates higher perceived stigma related to PrEP. The PrEP Stigma will be assessed at Baseline, Weeks 4, 8, and 12.
Time Frame: Baseline and up to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 2 Standard of Care | Part 2 Mini-app
Number analyzed (Participants) | 21 | 43
score on a scale
  Baseline to Week 4 | 0.06 (0.32) | -0.02 (0.69)
  Baseline to Week 8 | 0.23 (0.79) | 0.09 (0.72)
  Baseline to Week 12 | 0.02 (0.44) | 0.03 (0.72)
Statistical Analysis 1: Comparison: Part 2 Standard of Care vs Part 2 Mini-app; The comparison was made using data measured at Week 12; Test type: Superiority; p = 0.85, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Number of Participants Who Ordered At-home HIV/Syphilis Tests
Description: Number of participants who ordered at-home HIV/syphilis tests through the mini-app based on the study record. Values range from 0 to greater than 0. Higher indicates higher frequency of participants who ordered HIV/syphilis tests completed through the study.
Time Frame: 12 weeks
Population: This outcome is only applicable to the participants in the Part 2 mini-app arm who had access to the At-home HIV/syphilis tests per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Standard of Care | Part 2 Mini-app
Number analyzed (Participants) | 0 | 46
Participants |  | 13

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through the end of the study, a total of approximately 12 to 16 weeks.
Arm/Group | Part 2 Standard of Care | Part 2 Mini-app
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/46
Other Adverse Events (participants affected / at risk) | 0/24 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/56/NCT04426656/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT04426656/ICF_001.pdf